CLINICAL TRIAL: NCT05583097
Title: Selective Ultrasound Guided Cytology Using EU-TIRADS Versus Non-selective Ultrasound Guided Cytology for Diagnosing Thyroid Cancer
Brief Title: The Ultracyt Study - is EU-TIRADS Useful in Selecting Nodules for Fine Needle Aspiration Cytology?
Acronym: Ultracyt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Ultracyt 1.0
Record Dates: First submitted 2022-10-10; First posted 2022-10-17 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Thyroid Cancer; Thyroid Nodule
Keywords: Ultrasonography; Cytology; Thyroid Cancer; Thyroid Nodule; Diagnostics
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule

STUDY DESIGN:
Intervention Model Description: Randomization 1:1 in blocks of 10.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Selective cytology according to EU-TIRADS (No Intervention): All thyroid nodules are evaluated according to EU-TIRADS and cytology is performed according to EU-TIRADS criteria.
- Non-selective cytology (Active Comparator): All thyroid nodules are evaluated according to EU-TIRADS and cytology is performed on all nodules >1 cm. Cytology will also be performed on EU-TIRADS 5-nodules measuring between 0.5 and 1 cm.
  Interventions: Diagnostic Test: Non-selective cytology

INTERVENTIONS:
Diagnostic Test: Non-selective cytology — All noduleas are evaluated according to EU-TIRADS. Cytology performed on all nodules larger than 1 cm regardless of ultrasonographic features. Nodules 1 cm or smaller evaluated as EU-TIRADS 5 undergo cytologic examination if possible.
  Arms: Non-selective cytology

SUMMARY:
This is a randomized study evaluating selective fine-needle aspiration cytology based on structured ultrasound using EU-TIRADS versus non-selective ultrasound guided cytology. Primary outcome is frequency of suspicious cytology (Bethesda III-VI) which is expected to be higher in the selective group compared to the non-selective group. Secondary outcome is the frequency of malignancy which is expected to be equal in both groups. However, the investigators do not expect to reach statistical significance for the secondary outcome according to power calculations.

DETAILED DESCRIPTION:
Thyroid nodules are common in the population, and the reported incidence of thyroid cancer is increasing in most parts of the world. Palpable thyroid nodules are reported in 4-5 per cent of the population, of which 5-10 per cent are malignant. The reported incidence of thyroid nodules on ultrasound is higher.

EU-TIRADS has been shown in retrospective cohort studies to accurately stratify thyroid nodules with respect to risk of thyroid cancer. EU-TIRADS has been used in Western Sweden since 2017 and in 2021 it was implemented in the Swedish National Guidelines for thyroid cancer. To the knowledge of the investigators, no randomized controlled study has been carried out validating EU-TIRADS. This multicenter regional study aims to investigate the safety of using selective cytology using EU-TIRADS. Primary outcome is the result of cytology suspicious of thyroid cancer. In the selective group, low risk nodules will not undergo cytology and therefore the frequency of cytologically suspicious nodules (Bethesda III-VI) is expected to be higher in this group.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to ultrasonography of the thyroid due to goiter symtoms or positive findings on FDG-PET

Exclusion Criteria:

* Patients previously examined with ultrasonography of the thyroid
* Patients who have previously undergone thyroid surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency of suspicious cytology (Bethesda III-VI) in each arm. | Through study completion, up to 18 months.
  Fewer nodules in the selective cytology group will most likely undergo fine needle aspiration cytology (FNAC). However, since ultrasonographically benign nodules will not undergo FNAC the frequency of Bethesda III-VI is expected to be higher in the selective cytology group.

SECONDARY OUTCOMES:
Frequency of malignancy | Through study completion, up to 18 months.
  The frequency of malignancy is expected to be similar in both groups. Only patients undergoing surgery will be included in this analysis. The investigators do not expect to find statistical significance according to power calculations.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Muth, MD, PhD, Principal Investigator — Göteborg University
Locations (1):
- Department of radiology, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be made available including data, study protocol, statistical analysis plan and informed consent form.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available from six months to ten years after last patient inclusion in the study.
Access Criteria: Upon reasonable request data from the study will be made available by email to dr Jakob Dahlberg (jakob.dahlberg@vgregion.se) or dr Andreas Muth (andreas.muth@vgregion.se).
URL: https://www.gu.se/forskning/tyreoideacancer

REFERENCES:
- [Background] Russ G, Bonnema SJ, Erdogan MF, Durante C, Ngu R, Leenhardt L. European Thyroid Association Guidelines for Ultrasound Malignancy Risk Stratification of Thyroid Nodules in Adults: The EU-TIRADS. Eur Thyroid J. 2017 Sep;6(5):225-237. doi: 10.1159/000478927. Epub 2017 Aug 8. PMID 29167761
- [Background] Cibas ES, Ali SZ. The 2017 Bethesda System for Reporting Thyroid Cytopathology. Thyroid. 2017 Nov;27(11):1341-1346. doi: 10.1089/thy.2017.0500. PMID 29091573
- See also: EU-TIRADS description — https://pubmed.ncbi.nlm.nih.gov/29167761/
- See also: Updated description of the Bethesda system — https://pubmed.ncbi.nlm.nih.gov/29091573/
- Available data/document: Study Protocol — https://www.gu.se/forskning/tyreoideacancer